CLINICAL TRIAL: NCT03769051
Title: Study on The Oral Immune Tolerance of CMPA Infants Using Amino Acid Formula
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20180402 v1.3
Record Dates: First submitted 2018-11-01; First posted 2018-12-07 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2018-11

CONDITIONS: Cow's Milk Protein Allergy
Keywords: Cow's Milk Protein allergy; Open Food Challenge test; Immune Tolerance; Amino Acid Formula
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main purpose of this study was to observe the effect of amino acid formula on infants with cow's milk protein allergy; to evaluate the role of food avoidance and Open Food Challenge test in the diagnosis of infants with cow's milk protein allergy; to observe the allergic process in infants with cow's milk protein allergy and to explore the criteria for diagnosis and treatment.

DETAILED DESCRIPTION:
This is a multi-center, prospective cohort study. This study plans to recruit 200 subjects. The suitable subject will be enrolled and there are seven visits through the 6-month study. Efficacy parameters are the positive incidence of open food challenge test, growth and development index (Weight, Height, Head circumference;), and the improvement of CMPA symptoms (such as SCORAD, gastrointestinal tract, respiratory, comfort scores).

ELIGIBILITY:
Inclusion Criteria:

* Age: 0 to 6 months;
* Subject with cow's milk protein allergy (any clinical signs or symptoms of the skin, gastrointestinal tract, respiratory tract or comfortable tract)
* Unable to breastfeed;
* Vital signs are stable;
* Legal guardian has signed the informed consent.

Exclusion Criteria:

* Subject with congenital and hereditary metabolic diseases;
* Digestive tract obstruction;
* Subject with immunodeficiency diseases;
* Subject who is allergic to known components of amino acid formula powder;
* The investigator judges it is not suitable for the subject to participate in this study.

Ages: 1 Day to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Cow's milk protein allergy infants in 0~6 months
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2015-06-20 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Negative rate of open food challenge test | From baseline to AAF feeding for 6 months
  Negative rate =The subjects number with negative results of open food challenge test/total subject number with open food challenge test Unit:% Negative rate range: 0-100% High negative rate indicates the immune tolerance of CMPA infant using AAF

SECONDARY OUTCOMES:
WAZ(weight for age Z score) | From baseline to AAF feeding for 6 months
  Z-scores of anthropometric parameters from baseline on weight=Average(The difference between the measured infant weight and the reference infant weight of the same age and sex/the reference infant weight standard deviation) The increase of WAZ indicated that AAF could promote growth and development.
HAZ(height for age Z score) | From baseline until AAF feeding for 6 months
  Z-scores of anthropometric parameters from baseline on height=Average(The difference between the measured infant height and the reference infant height of the same age and sex/the reference infant height standard deviation) The increase of HAZ indicated that AAF could promote growth and development.
HCAZ(head circumference for age Z score) | From baseline to AAF feeding for 6 months
  Z-scores of anthropometric parameters from baseline on head circumference=Average(The difference between the measured infant head circumference and the reference infant head circumference of the same age and sex/the reference infant head circumference standard deviation) The increase of HCAZ indicated that AAF could promote growth and development.
SCORAD score | From baseline to AAF feeding for 6 months
  An SCORAD evaluation scale was evaluated by the investigator at each visit
Gastrointestinal symptom score | From baseline to AAF feeding for 6 months
  An Gastrointestinal symptom evaluation scale was evaluated by the investigator at each visit
Respiratory symptom score | From baseline to AAF feeding for 6 months
  An Respiratory symptom evaluation scale was evaluated by the investigator at each visit
Comfort symptom score | From baseline to AAF feeding for 6 months
  An Comfort symptom evaluation scale was evaluated by the investigator at each visit

CONTACTS AND LOCATIONS:
Overall Officials: Juan Zhang, Study Director — Colleague

IPD SHARING:
Plan to Share IPD: Undecided